CLINICAL TRIAL: NCT07374835
Title: BMI Stratified Management Based on Meridian-Lymph Axis Theory for Lower Extremity Lymphedema in Patients After Gynecologic Cancer Surgery
Brief Title: BMI Stratified Management Based on Meridian-Lymph Axis Theory for Lower Extremity Lymphedema After Gynecologic Cancer Surgery
Acronym: MLA-BMI-LLE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Zhang (Other)
Responsible Party: Sponsor-Investigator, Hong Zhang, Associate Chief Nurse, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB202512073
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Lower Extremity Lymphedema After Gynecologic Cancer Surgery
Keywords: Gynecologic Cancer Surgery; Lower Extremity Lymphedema; BMI Stratified Management; Meridian-Lymph Axis Theory

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMI Stratified Management Group (Experimental): Participants receive personalized management based on BMI, combining meridian conditioning and lymphatic circulation interventions.
  Interventions: Other: Meridian-Lymph Axis Based BMI Stratified Management
- Routine Care Control Group (Other): Participants receive standard lymphatic edema care (e.g., compression garments, basic exercise guidance).
  Interventions: Other: Routine Lymphatic Edema Care

INTERVENTIONS:
Other: Meridian-Lymph Axis Based BMI Stratified Management — Personalized interventions including meridian point stimulation, manual lymphatic drainage, and pressure care, stratified by participant BMI.
  Arms: BMI Stratified Management Group
Other: Routine Lymphatic Edema Care — Standard care including compression garment use, limb elevation, and basic exercise guidance.
  Arms: Routine Care Control Group

SUMMARY:
This study aims to investigate the impact of a BMI-stratified intervention program based on the meridian-lymphatic axis theory on the incidence of lower extremity lymphedema in postoperative patients with gynecological malignant tumors at 1 month, 3 months, and 6 months, and to validate the precision and effectiveness of this program compared to traditional CDT. Primary objectives: to evaluate the effects of this program on reducing the incidence of lymphedema, alleviating lymphedema-related symptoms (assessed via GCLQ score), improving patients' quality of life (assessed via LLQoL score), and enhancing patients' self-management behaviors.

ELIGIBILITY:
Inclusion Criteria:Female patients aged 18-75 years who have undergone gynecologic cancer surgery (including hysterectomy, oophorectomy, or lymphadenectomy).

Diagnosed with lower extremity lymphedema (stage I-II) within 6 months to 2 years post-surgery, confirmed by circumferential measurement.

BMI between 18.5 and 35.0 kg/m². Able to understand and sign the informed consent form, and comply with the intervention and follow-up schedule.

No history of severe cardiovascular, renal, or hepatic dysfunction that would interfere with study participation.

-

Exclusion Criteria:Patients with lower extremity lymphedema caused by other etiologies (e.g., trauma, infection, or congenital lymphedema).

History of lower extremity surgery or fracture within 3 months prior to enrollment.

Active infection or skin ulceration in the affected lower extremity. Participation in other clinical trials involving lymphedema interventions within the past 3 months.

Pregnancy or lactation during the study period. Inability to complete the intervention or follow-up due to cognitive or mobility impairment.

-

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Lower Extremity Lymphedema Volume (Measured by Circumferential Method) | Baseline (before intervention), 12 weeks after intervention initiation
  Limb volume change will be calculated using circumferential measurements of the lower extremity (ankle, calf, thigh) to quantify the reduction in lymphedema severity after intervention.
Change in Lower Extremity Lymphedema Volume (measured by circumferential measurement) from baseline to 12 weeks after intervention | Baseline, 12 weeks
  Limb volume change will be calculated using circumferential measurements of the lower extremity to assess the efficacy of the intervention in reducing lymphedema.

SECONDARY OUTCOMES:
Change in Limb Function Score (using the Lymphoedema Functioning, Disability and Health Questionnaire, LYMPH-Q) from baseline to 12 weeks | baseline to 12 weeks
Change in Quality of Life Score (using the European Organization for Research and Treatment of Cancer QLQ-C30) from baseline to 12 weeks | baseline to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-10-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT07374835/SAP_000.pdf